CLINICAL TRIAL: NCT02114398
Title: Physiotherapy Efficiency With Caycedian Sophrology on Child Asthma: Randomized, Controlled Study
Brief Title: Physiotherapy Efficiency on Child Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 9162
Record Dates: First submitted 2014-02-26; First posted 2014-04-15 (Estimated); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Child; Asthma Crisis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- usual treatment (Experimental): usual treatment
  Interventions: Other: usual treatment
- usual treatment + sophrology (Experimental): usual treatment + sophrology
  Interventions: Other: usual treatment + sophrology

INTERVENTIONS:
Other: usual treatment — usual treatment
  Arms: usual treatment
Other: usual treatment + sophrology — usual treatment + sophrology
  Arms: usual treatment + sophrology

SUMMARY:
The study aim is to compare usual asthma crisis treatment of hospitalized children with usual treatment associated to sophrology.

ELIGIBILITY:
Inclusion Criteria:

* child (6 to 17 years old)
* hospitalized in pediatric unit for asthma crisis

Exclusion Criteria:

* patient who can't participate because of his healthcare (resuscitation...)
* impossibility to measure Peak Expiratory Flow (PEF)

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2013-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Peak Expiratory Flow (PEF) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Pascal AMEDRO, MD, PhD, Principal Investigator — UH Montpellier
Locations (1):
- Pediatric and Congenital Cardiology and Pulmonology Department, Arnaud De Villeneuve University Hospital, Montpellier, France

REFERENCES:
- [Result] Romieu H, Charbonnier F, Janka D, Douillard A, Macioce V, Lavastre K, Abassi H, Renoux MC, Mura T, Amedro P. Efficiency of physiotherapy with Caycedian Sophrology on children with asthma: A randomized controlled trial. Pediatr Pulmonol. 2018 May;53(5):559-566. doi: 10.1002/ppul.23982. Epub 2018 Mar 1. PMID 29493875